CLINICAL TRIAL: NCT00868725
Title: Detecting Lesions in the Oral Cavity With Thermal Imaging
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Prof. Arie Orenstein , Director Advanced Technologies Center, Sheba Medical Center
Other Study IDs: SHEBA-09-6870-AO-CTIL
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-09

CONDITIONS: Carcinoma, Squamous Cell
Keywords: oral cavity; carcinoma; thermal imaging
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- possible oral cancer: Patients reporting for oral cavity examination with the possibility or certainty of oral lesions
  Interventions: Other: no intervention, observation only

INTERVENTIONS:
Other: no intervention, observation only — Oral cavity will be imaged by a thermal camera.

SUMMARY:
Previous studies indicate that there are significant differences in the temperature of tumors and normal, adjacent tissues. The present study will test this hypothesis for lesions in the oral cavity. Thermal images of the oral cavities of patients, undergoing examination in the Department of Oral and Maxillofacial Surgery of Sheba hospital, will be compared to the diagnoses of the examining doctors. The results, apart from enhancing the delineation of oral cavity tumors, may help the decision to develop miniature thermal cameras to scan thermally, the GI tract.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed in the Department of Oral and Maxillofacial Surgery as suffering from malignant or possibly malignant lesions.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients reporting for oral cavity examination under the possibility of presenting with oral cavity lesions
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Ability of a thermal camera to detect and delineate tumors in the oral cavity | during and immediately after the examination

CONTACTS AND LOCATIONS:
Overall Officials: Arie Orenstein, Prof., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Stefanadis C, Chrysohoou C, Panagiotakos DB, Passalidou E, Katsi V, Polychronopoulos V, Toutouzas PK. Temperature differences are associated with malignancy on lung lesions: a clinical study. BMC Cancer. 2003 Jan 6;3:1. doi: 10.1186/1471-2407-3-1. Epub 2003 Jan 6. PMID 12515579